CLINICAL TRIAL: NCT01062256
Title: A Methodology Study to Assess Cough Counts in Subjects With Acute Upper Respiratory Tract Infections
Brief Title: Study of Count Coughs in Subjects With Acute Upper Respiratory Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GG-09-06; B4361001
Record Dates: First submitted 2010-02-01; First posted 2010-02-04 (Estimated); Results first posted 2011-03-04 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Infection
Keywords: Cough assessment in upper respiratory infection; guaifenesin; honey
MeSH Terms: conditions — Infections | interventions — Guaifenesin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Guaifenesin (Experimental): Guaifenesin
  Interventions: Drug: Guaifenesin
- Buckwheat Honey (Experimental): Buckwheat Honey
  Interventions: Other: Buckwheat Honey

INTERVENTIONS:
Drug: Placebo — One placebo tablet administered orally as a single dose
  Arms: Placebo
Drug: Guaifenesin — One 400 mg immediate release tablet administered orally as a single dose
  Arms: Guaifenesin
Other: Buckwheat Honey — 10 mL administered orally as a single dose
  Arms: Buckwheat Honey

SUMMARY:
The objectives of this study are: a) to assess the feasibility and sensitivity of manually count cough bouts over a 4-hour period; b) to assess the effects of buckwheat honey and guaifenesin 400 mg immediate release tablets compared to placebo on the frequency and severity of acute cough due to upper respiratory tract infection and c) to evaluate the correlation between cough bout frequency and subjective assessments of cough severity. The hypotheses to be tested is that 10 ml of buckwheat honey and 400 mg of immediate release guaifenesin will significantly reduce the frequency and severity of cough compared to placebo over a 4-hour evaluation period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at least 18 years of age and in generally good health who are experiencing an acute upper respiratory infection of 10 days or less in duration;
* Subjects currently have acute cough self-rated as at least moderate due to an acute Upper Respiratory Infection (URTI) (i.e., cold or flu) as established by a study physician, nurse practitioner, or physician's assistant;
* Subjects who have > 5 cough bouts during the 30 minute baseline assessment period

Exclusion Criteria:

* Subjects who have acute, subchronic, or chronic cough due to any condition other than a URTI as established by the Investigator, nurse practitioner, or physician's assistant, in accordance with the American College of Chest Physicians (ACCP) Guidelines for Diagnosis and Management of Cough. Special attention should be paid to highly prevalent conditions commonly presenting with cough such as asthma, Chronic Obstructive Pulmonary Disease (COPD), and Gastroesophageal Reflux Disease (GERD) (N.B. Subjects with exercise-induced asthma may be eligible for the study as long as they have not experienced an episode of asthma within 24 hours of enrollment)
* In the opinion of a study physician, nurse practitioner, or physician's assistant, subjects with sinusitis or who have a history of (within the past 2 years) frequent clinically significant sinusitis;
* Subjects with a history (within the last 3 years) of alcohol abuse (i.e., consuming greater than or equal to 3 alcoholic drinks/day on a regular basis) or substance abuse (i.e., ingesting/smoking marijuana more than once a week at any time during the past 6 months or using any other recreational drug more than once during the past 6 months). (Note: One "drink" of alcohol=1 oz. liquor, 6 oz wine, 12 oz. beer.);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Lexington, Kentucky

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=GG-09-06&StudyName=Study%20of%20Count%20Coughs%20in%20Subjects%20with%20Acute%20Upper%20Respiratory%20Tract%20Infections%20%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants stratified by gender and time of dosing (before or at 3:00 pm versus after 3:00 pm).
Groups:
- Buckwheat Honey: 10 milliliters (mL) administered orally as a single dose
- Guaifenesin: One 400 milligrams (mg) immediate release tablet administered orally as a single dose
Period: Overall Study
Arm/Group | Placebo | Buckwheat Honey | Guaifenesin
Started | 55 | 103 | 107
Completed | 52 | 96 | 103
Not Completed | 3 | 7 | 4
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Ineligible | 1 | 4 | 3
Not completed — Administrative | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Buckwheat Honey | Guaifenesin | Total
Number analyzed (Participants) | 55 | 103 | 107 | 265
Age Continuous [Mean (Standard Deviation); unit: years] | 29.9 (9.5) | 33.5 (11.2) | 32.4 (11.1) | 32.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 62 | 64 | 159
  Male | 22 | 41 | 43 | 106

OUTCOME MEASURES:

1. Primary Outcome: Number of Cough Bouts Over 4-hour Postdose Period
Description: Cough bouts defined as one or several cough sounds occurring after one inspiration (one explosive bout between inspiration and expiration). Audio recordings made of participants during 4-hour period after dosing. Based on audio recordings, a trained cough counter counted and recorded the number of cough bouts.
Time Frame: 0 to 4 hours postdose
Population: Intent-to-Treat (ITT) Population: all randomized participants who provided baseline cough counts and were dosed with study product.
Measure: Mean (Standard Deviation); unit: Cough bouts
Arm/Group | Placebo | Buckwheat Honey | Guaifenesin
Number analyzed (Participants) | 54 | 102 | 107
Cough bouts | 139.6 (140.6) | 131.3 (138.8) | 126.4 (126.1)
Statistical Analysis 1: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of number of cough bouts over 4-hour postdose period; Test type: Superiority or Other; p = 0.216, Poisson regression model — p-values calculated from Poisson regression model with treatment, gender, time stratum (dosing before or at 3:00 pm, or after 3:00 pm), site, and baseline of cough bouts terms with log(exposure time) as the offset parameter; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.64 to 1.10]
Statistical Analysis 2: Comparison: Placebo vs Guaifenesin; Pairwise comparison of number of cough bouts over 4-hour postdose period; Test type: Superiority or Other; p = 0.513, Poisson regression model — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.72 to 1.18]
Statistical Analysis 3: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of number of cough bouts over 4-hour postdose period; Test type: Superiority or Other; p = 0.459, Poisson regression model — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.87 to 1.38]

2. Secondary Outcome: Number of Cough Bouts Over 2-hour Postdose Period
Description: Cough bouts defined as one or several cough sounds occurring after one inspiration (one explosive bout between inspiration and expiration). Audio recordings made of participants during first 2 hours postdose. Based on audio recordings, a trained cough counter counted and recorded the number of cough bouts.
Time Frame: 0 to 2 hours postdose
Population: ITT
Measure: Mean (Standard Deviation); unit: cough bouts
Arm/Group | Placebo | Buckwheat Honey | Guaifenesin
Number analyzed (Participants) | 54 | 102 | 107
cough bouts | 83.8 (81.9) | 79.8 (81.8) | 75.0 (71.9)
Statistical Analysis 1: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of number of cough bouts over 2-hour postdose period; Test type: Superiority or Other; p = 0.195, Poisson regression model — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.65 to 1.09]
Statistical Analysis 2: Comparison: Placebo vs Guaifenesin; Pairwise comparison of number of cough bouts over 2-hour postdose period; Test type: Superiority or Other; p = 0.438, Poisson regression model — p-values calculated from Poisson regression model with treatment, gender, time stratum (dosing before or at 3:00 pm, or after 3:00 pm), site and baseline of cough bouts terms with log(exposure time)as the offset parameter; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.71 to 1.16]
Statistical Analysis 3: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of number of cough bouts over 2-hour postdose period; Test type: Superiority or Other; p = 0.497, Poisson regression model — [p-value comment as in outcome 2, analysis 2]; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.87 to 1.34]

3. Secondary Outcome: Number of Cough Bouts Within Each 15-minute Time Interval Postdose
Description: Cough bouts defined as one or several cough sounds occurring after one inspiration (one explosive bout between inspiration and expiration). Audio recordings made of participants during 4-hour (240-minute) period after dosing. Based on audio recordings, a trained cough counter counted and recorded the number of cough bouts in 15 minute intervals.
Time Frame: every 15 minutes postdose up to 240 minutes postdose
Population: ITT
Measure: Mean (Standard Deviation); unit: cough bouts
Arm/Group | Placebo | Buckwheat Honey | Guaifenesin
Number analyzed (Participants) | 54 | 102 | 107
cough bouts
  15 minutes | 14.9 (16.8) | 14.5 (14.3) | 14.2 (12.4)
  30 minutes | 12.4 (13.0) | 10.9 (10.9) | 11.0 (11.0)
  45 minutes | 11.5 (11.4) | 10.6 (12.2) | 9.5 (9.5)
  60 minutes | 10.1 (10.5) | 9.6 (10.0) | 8.7 (9.5)
  75 minutes | 8.1 (9.6) | 8.7 (10.0) | 8.2 (8.6)
  90 minutes | 9.4 (10.3) | 8.7 (10.5) | 8.0 (9.1)
  105 minutes | 9.6 (10.0) | 8.6 (9.9) | 7.9 (9.1)
  120 minutes | 8.3 (7.9) | 8.4 (9.8) | 7.9 (9.3)
  135 minutes | 6.8 (7.0) | 7.2 (9.6) | 6.6 (8.1)
  150 minutes | 7.9 (8.6) | 7.1 (8.7) | 6.8 (7.8)
  165 minutes | 7.7 (8.6) | 7.0 (8.3) | 7.0 (8.2)
  180 minutes | 6.5 (7.1) | 6.9 (8.3) | 6.9 (8.0)
  195 minutes | 6.1 (7.8) | 6.3 (8.4) | 5.9 (6.8)
  210 minutes | 6.8 (7.8) | 5.7 (7.6) | 6.3 (7.6)
  225 minutes | 7.2 (8.9) | 5.8 (7.5) | 6.0 (7.6)
  240 minutes | 7.1 (9.1) | 5.9 (8.7) | 6.3 (8.5)
Statistical Analysis 1: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of the number of cough bouts within 15 minutes postdose; Test type: Superiority or Other; p = 0.250, Poisson regression model — p-values from Poisson regression model with treatment, gender, time stratum (dosing before or at 3:00 pm, or after 3:00 pm), site, and baseline of cough bouts terms with log(exposure time); Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.64 to 1.12]
Statistical Analysis 2: Comparison: Placebo vs Guaifenesin; Pairwise comparison of the number of cough bouts within 15 minutes postdose; Test type: Superiority or Other; p = 0.802, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.75 to 1.25]
Statistical Analysis 3: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of the number of cough bouts within 15 minutes postdose; Test type: Superiority or Other; p = 0.188, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.94 to 1.39]
Statistical Analysis 4: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of the number of cough bouts between 15 and 30 minutes postdose; Test type: Superiority or Other; p = 0.091, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.58 to 1.04]
Statistical Analysis 5: Comparison: Placebo vs Guaifenesin; Pairwise comparison of the number of cough bouts between 15 and 30 minutes postdose; Test type: Superiority or Other; p = 0.465, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.69 to 1.19]
Statistical Analysis 6: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of the number of cough bouts between 15 and 30 minutes postdose; Test type: Superiority or Other; p = 0.207, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.92 to 1.46]
Statistical Analysis 7: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of the number of cough bouts between 30 and 45 minutes postdose; Test type: Superiority or Other; p = 0.122, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.62 to 1.06]
Statistical Analysis 8: Comparison: Placebo vs Guaifenesin; Pairwise comparison of the number of cough bouts between 30 and 45 minutes postdose; Test type: Superiority or Other; p = 0.165, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.66 to 1.07]
Statistical Analysis 9: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of the number of cough bouts between 30 and 45 minutes postdose; Test type: Superiority or Other; p = 0.711, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.83 to 1.32]
Statistical Analysis 10: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of the number of cough bouts between 45 and 60 minutes postdose; Test type: Superiority or Other; p = 0.215, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.64 to 1.11]
Statistical Analysis 11: Comparison: Placebo vs Guaifenesin; Pairwise comparison of the number of cough bouts between 45 and 60 minutes postdose; Test type: Superiority or Other; p = 0.367, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.67 to 1.16]
Statistical Analysis 12: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of the number of cough bouts between 45 and 60 minutes postdose; Test type: Superiority or Other; p = 0.687, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.82 to 1.35]
Statistical Analysis 13: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of the number of cough bouts between 60 and 75 minutes postdose; Test type: Superiority or Other; p = 0.730, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.67 to 1.32]
Statistical Analysis 14: Comparison: Placebo vs Guaifenesin; Pairwise comparison of the number of cough bouts between 60 and 75 minutes postdose; Test type: Superiority or Other; p = 0.923, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.74 to 1.39]
Statistical Analysis 15: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of the number of cough bouts between 60 and 75 minutes postdose; Test type: Superiority or Other; p = 0.573, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.83 to 1.40]
Statistical Analysis 16: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of the number of cough bouts between 75 and 90 minutes postdose; Test type: Superiority or Other; p = 0.289, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.61 to 1.16]
Statistical Analysis 17: Comparison: Placebo vs Guaifenesin; Pairwise comparison of the number of cough bouts between 75 and 90 minutes postdose; Test type: Superiority or Other; p = 0.379, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.64 to 1.18]
Statistical Analysis 18: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of the number of cough bouts between 75 and 90 minutes postdose; Test type: Superiority or Other; p = 0.785, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.79 to 1.37]
Statistical Analysis 19: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of the number of cough bouts between 90 and 105 minutes postdose; Test type: Superiority or Other; p = 0.194, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.60 to 1.11]
Statistical Analysis 20: Comparison: Placebo vs Guaifenesin; Pairwise comparison of the number of cough bouts between 90 and 105 minutes postdose; Test type: Superiority or Other; p = 0.212, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.62 to 1.11]
Statistical Analysis 21: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of the number of cough bouts between 90 and 105 minutes postdose; Test type: Superiority or Other; p = 0.901, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.77 to 1.34]
Statistical Analysis 22: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of the number of cough bouts between 105 and 120 minutes postdose; Test type: Superiority or Other; p = 0.600, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.70 to 1.23]
Statistical Analysis 23: Comparison: Placebo vs Guaifenesin; Pairwise comparison of the number of cough bouts between 105 and 120 minutes postdose; Test type: Superiority or Other; p = 0.853, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.74 to 1.29]
Statistical Analysis 24: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of the number of cough bouts between 105 and 120 minutes postdose; Test type: Superiority or Other; p = 0.736, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.79 to 1.39]
Statistical Analysis 25: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of the number of cough bouts between 120 and 135 minutes postdose; Test type: Superiority or Other; p = 0.744, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.70 to 1.30]
Statistical Analysis 26: Comparison: Placebo vs Guaifenesin; Pairwise comparison of the number of cough bouts between 120 and 135 minutes postdose; Test type: Superiority or Other; p = 0.904, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.72 to 1.33]
Statistical Analysis 27: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of the number of cough bouts between 120 and 135 minutes postdose; Test type: Superiority or Other; p = 0.828, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.77 to 1.39]
Statistical Analysis 28: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of the number of cough bouts between 135 and 150 minutes postdose; Test type: Superiority or Other; p = 0.147, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.59 to 1.08]
Statistical Analysis 29: Comparison: Placebo vs Guaifenesin; Pairwise comparison of the number of cough bouts between 135 and 150 minutes postdose; Test type: Superiority or Other; p = 0.345, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.65 to 1.16]
Statistical Analysis 30: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of the number of cough bouts between 135 and 150 minutes postdose; Test type: Superiority or Other; p = 0.532, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.83 to 1.44]
Statistical Analysis 31: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of the number of cough bouts between 150 and 165 minutes postdose; Test type: Superiority or Other; p = 0.261, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.61 to 1.15]
Statistical Analysis 32: Comparison: Placebo vs Guaifenesin; Pairwise comparison of the number of cough bouts between 150 and 165 minutes postdose; Test type: Superiority or Other; p = 0.601, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.69 to 1.24]
Statistical Analysis 33: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of the number of cough bouts between 150 and 165 minutes postdose; Test type: Superiority or Other; p = 0.470, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.84 to 1.47]
Statistical Analysis 34: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of the number of cough bouts between 165 and 180 minutes postdose; Test type: Superiority or Other; p = 0.834, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.71 to 1.32]
Statistical Analysis 35: Comparison: Placebo vs Guaifenesin; Pairwise comparison of the number of cough bouts between 165 and 180 minutes postdose; Test type: Superiority or Other; p = 0.628, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.81 to 1.43]
Statistical Analysis 36: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of the number of cough bouts between 165 and 180 minutes postdose; Test type: Superiority or Other; p = 0.481, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.83 to 1.48]
Statistical Analysis 37: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of the number of cough bouts between 180 and 195 minutes postdose; Test type: Superiority or Other; p = 0.749, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.65 to 1.37]
Statistical Analysis 38: Comparison: Placebo vs Guaifenesin; Pairwise comparison of the number of cough bouts between 180 and 195 minutes postdose; Test type: Superiority or Other; p = 0.857, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.70 to 1.35]
Statistical Analysis 39: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of the number of cough bouts between 180 and 195 minutes postdose; Test type: Superiority or Other; p = 0.847, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.76 to 1.41]
Statistical Analysis 40: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of the number of cough bouts between 195 and 210 minutes postdose; Test type: Superiority or Other; p = 0.146, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.54 to 1.09]
Statistical Analysis 41: Comparison: Placebo vs Guaifenesin; Pairwise comparison of the number of cough bouts between 195 and 210 minutes postdose; Test type: Superiority or Other; p = 0.702, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.69 to 1.29]
Statistical Analysis 42: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of the number of cough bouts between 195 and 210 minutes postdose; Test type: Superiority or Other; p = 0.228, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.88 to 1.69]
Statistical Analysis 43: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of the number of cough bouts between 210 and 225 minutes postdose; Test type: Superiority or Other; p = 0.130, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.51 to 1.09]
Statistical Analysis 44: Comparison: Placebo vs Guaifenesin; Pairwise comparison of the number of cough bouts between 210 and 225 minutes postdose; Test type: Superiority or Other; p = 0.371, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.60 to 1.21]
Statistical Analysis 45: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of the number of cough bouts between 210 and 225 minutes postdose; Test type: Superiority or Other; p = 0.430, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.82 to 1.58]
Statistical Analysis 46: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of the number of cough bouts between 225 and 240 minutes postdose; Test type: Superiority or Other; p = 0.177, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.51 to 1.13]
Statistical Analysis 47: Comparison: Placebo vs Guaifenesin; Pairwise comparison of the number of cough bouts between 225 and 240 minutes postdose; Test type: Superiority or Other; p = 0.580, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.64 to 1.28]
Statistical Analysis 48: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of the number of cough bouts between 225 and 240 minutes postdose; Test type: Superiority or Other; p = 0.333, Poisson regression model — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.84 to 1.70]

4. Secondary Outcome: Change From Baseline in Cough Severity Scale
Description: Participant's self-assessment of cough severity using a 4-point categorical scale (0 = none; no cough present, 1 = mild; cough present but with minimal awareness, easily tolerated, 2 = moderate; cough definitely present and bothersome, but tolerable, or 3 = severe; cough was hard to tolerate; may have caused interference with daily activities and sleeping). Change from baseline derived by subtracting post baseline cough severity from baseline cough severity. Change from baseline values could have ranged from -1.0 to 3.0 with higher values indicative of greater improvement.
Time Frame: 1, 2, 3, and 4 hours postdose
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Buckwheat Honey | Guaifenesin
Number analyzed (Participants) | 54 | 102 | 107
units on a scale
  1 hour postdose | 0.4 (0.5) | 0.5 (0.6) | 0.3 (0.5)
  2 hours postdose | 0.6 (0.6) | 0.7 (0.6) | 0.6 (0.6)
  3 hours postdose | 0.8 (0.6) | 1.0 (0.6) | 0.8 (0.7)
  4 hours postdose | 1.0 (0.7) | 1.1 (0.7) | 1.0 (0.7)
Statistical Analysis 1: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of change from baseline in cough severity at 1 hour postdose; Test type: Superiority or Other; p = 0.264, ANOVA — p-values from ANOVA model with treatment, gender, time stratum (dosing before or at 3:00 pm, or after 3:00 pm), and site terms; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.08 to 0.27]
Statistical Analysis 2: Comparison: Placebo vs Guaifenesin; Pairwise comparison of change from baseline in cough severity at 1 hour postdose; Test type: Superiority or Other; p = 0.737, ANOVA — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.20 to 0.14]
Statistical Analysis 3: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of change from baseline in cough severity at 1 hour postdose; Test type: Superiority or Other; p = 0.078, ANOVA — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.27 to 0.01]
Statistical Analysis 4: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of change from baseline in cough severity at 2 hour postdose; Test type: Superiority or Other; p = 0.125, ANOVA — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.04 to 0.36]
Statistical Analysis 5: Comparison: Placebo vs Guaifenesin; Pairwise comparison of change from baseline in cough severity at 2 hour postdose; Test type: Superiority or Other; p = 0.688, ANOVA — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.16 to 0.24]
Statistical Analysis 6: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of change from baseline in cough severity at 2 hour postdose; Test type: Superiority or Other; p = 0.166, ANOVA — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.29 to 0.05]
Statistical Analysis 7: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of change from baseline in cough severity at 3 hour postdose; Test type: Superiority or Other; p = 0.233, ANOVA — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.09 to 0.35]
Statistical Analysis 8: Comparison: Placebo vs Guaifenesin; Pairwise comparison of change from baseline in cough severity at 3 hour postdose; Test type: Superiority or Other; p = 0.848, ANOVA — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.24 to 0.19]
Statistical Analysis 9: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of change from baseline in cough severity at 3 hour postdose; Test type: Superiority or Other; p = 0.093, ANOVA — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.33 to 0.03]
Statistical Analysis 10: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of change from baseline in cough severity at 4 hour postdose; Test type: Superiority or Other; p = 0.406, ANOVA — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.14 to 0.34]
Statistical Analysis 11: Comparison: Placebo vs Guaifenesin; Pairwise comparison of change from baseline in cough severity at 4 hour postdose; Test type: Superiority or Other; p = 0.991, ANOVA — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.24 to 0.24]
Statistical Analysis 12: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of change from baseline in cough severity at 4 hour postdose; Test type: Superiority or Other; p = 0.306, ANOVA — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.30 to 0.09]

5. Secondary Outcome: Number of Participants With Global Evaluation of Study Medication
Description: Participant-rated evaluation of study product; Participants responded to the following question:
  "How would you rate this product as a cough reliever?" 0=poor, 1=fair, 2=good, 3=very good, and 4=excellent
Time Frame: 4 hours postdose or early termination
Population: ITT
Measure: Number; unit: participants
Arm/Group | Placebo | Buckwheat Honey | Guaifenesin
Number analyzed (Participants) | 54 | 102 | 107
participants
  Poor | 5 | 9 | 11
  Fair | 18 | 28 | 39
  Good | 18 | 33 | 29
  Very Good | 10 | 22 | 23
  Excellent | 2 | 9 | 5
Statistical Analysis 1: Comparison: Placebo vs Buckwheat Honey; Pairwise comparison of global evaluation of study medication; Test type: Superiority or Other; p = 0.254, Cochran-Mantel-Haenszel — p-values from Cochran-Mantel-Haenszel test with modified ridit scores, controlling for gender, time stratum, and site; Goodman-Kruskal Gamma statistic = 0.15, 95% CI 2-sided [-0.09 to 0.39]
Statistical Analysis 2: Comparison: Placebo vs Guaifenesin; Pairwise comparison of global evaluation of study medication; Test type: Superiority or Other; p = 0.949, Cochran-Mantel-Haenszel — p-values from Cochran-Mantel-Haenszel test with modified ridit scores, controlling for gender, time stratum, and site; weighted Goodman-Kruskal Gamma statistic = -0.01, 95% CI 2-sided [-0.25 to 0.23]
Statistical Analysis 3: Comparison: Buckwheat Honey vs Guaifenesin; Pairwise comparison of global evaluation of study medication; Test type: Superiority or Other; p = 0.256, Cochran-Mantel-Haenszel — p-values from Cochran-Mantel-Haenszel test with modified ridit scores, controlling for gender, time stratum, and site; weighted Goodman-Kruskal Gamma statistic = -0.12, 95% CI 2-sided [-0.32 to 0.08]

6. Other Pre Specified Outcome: Number of Participant With Cough Severity
Description: Participant's self-assessment of cough severity using 4-point categorical scale (0 = none; no cough present, 1 = mild; cough present but with minimal awareness, easily tolerated, 2 = moderate; cough definitely present and bothersome, but tolerable, or 3 = severe; cough was hard to tolerate; may have caused interference with daily activities and sleeping). Participants were eligible for study if severity of cough at baseline was at least moderate.
Time Frame: Baseline
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Placebo | Buckwheat Honey | Guaifenesin
Number analyzed (Participants) | 54 | 102 | 107
Participants
  Moderate | 51 | 92 | 101
  Severe | 3 | 10 | 6

ADVERSE EVENTS:
Description: The same event may have appeared as both an adverse event (AE) and a serious adverse event (SAE). However, what was presented were distinct events. An event may have been categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Buckwheat Honey | Guaifenesin
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/103 | 0/107
Other Adverse Events (participants affected / at risk) | 3/55 | 3/103 | 4/107
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=55) | Buckwheat Honey (N=103) | Guaifenesin (N=107)
Chest discomfort (Cardiac disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Dry throat (Gastrointestinal disorders) | 0 | 1 | 0
Feeling jittery (General disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.